CLINICAL TRIAL: NCT06524167
Title: A Real-world Study of Adjuvant Radiotherapy in High Recurrence Risk Locally Advanced Thyroid Cancer
Brief Title: RW Study of Adjuvant Radiotherapy in Locally Advanced Thyroid Cancer
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Yu Wang, Chief of Head-neck surgery, Fudan University Shanghai Cancer Center, Fudan University
Other Study IDs: AREAL
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Radiotherapy, Adjuvant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adjuvant radiotherapy: Locally advanced recurrent high-risk thyroid cancer patients who had adjuvant radiotherapy.
  Interventions: Radiation: adjuvant radiotherapy

INTERVENTIONS:
Radiation: adjuvant radiotherapy — The patients would receive external radiation therapy within 6 weeks after surgery, using intensity-modulated radiation therapy (IMRT) or volume modulated radiation therapy (VMAT) techniques. 6MV-X-ray irradiation. Conventional segmented irradiation is used, once a day, five times a week, with a segmented dose of 2Gy per dose.

SUMMARY:
This study is a real-world study to observe the role of adjuvant radiotherapy in locally advanced recurrent high-risk thyroid cancer. The study included thyroid cancer that requires adjuvant radiotherapy to increase local control rate, excluding undifferentiated cancer. Local-regional recurrence free survival is the primary endpoint of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients voluntarily join this study and sign an informed consent form;
* Age: ≥ 14 years old,<80 years old, male or female not limited;
* Thyroid cancer diagnosed by histopathology, including differentiated thyroid cancer, medullary carcinoma, poorly differentiated carcinoma, etc;
* High risk of local late recurrence, meeting any of the following criteria:

  1. The surgery did not achieve R0 resection;
  2. After neoadjuvant therapy;
  3. Pathological types with poor prognosis, such as poorly differentiated cancer, CASTLE, etc;
  4. Thyroid cancer with obvious extracapsular invasion, invading important structures such as the esophagus, trachea, and recurrent laryngeal nerve, requiring adjuvant radiotherapy;
  5. For patients with distant metastasis, researchers need to determine the value of local treatment;
* The main organ functions are normal;
* Good compliance and cooperation with follow-up.

Exclusion Criteria:

* Untreated thyroid cancer or thyroid cancer that has only undergone surgical biopsy;
* Within 5 years or simultaneously suffering from other active malignant tumors. Cured local tumors, such as skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, prostate carcinoma in situ, cervical carcinoma in situ, breast carcinoma in situ, can be included in the group;
* Previously received radiation therapy for the head and neck area;
* Pregnant or lactating women;
* There are other physical illnesses that affect patients' ability to receive standard treatment;
* According to the researcher's judgment, there may be other factors that could force the subject to terminate the study midway, such as suffering from other serious illnesses (including mental illnesses) that require concurrent treatment, severe abnormal laboratory test values, family or social factors that may affect the subject's safety or the collection of trial data;
* Individuals with claustrophobia who are unable to undergo radiation therapy;
* Other patients deemed unsuitable for inclusion by the treating physician.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with high recurrence risk locally advanced thyroid cancer
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2031-06-30 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
LRRFS | 5 years
  Local-regional Recurrence Free Survival

SECONDARY OUTCOMES:
DCR | 5 years
  Disease Control Rate
PFS | 5 years
  Progression Free Survival
OS | 5 years
  Overall Survival
AE | 5 years
  Adverse Events
QoL | 5 years
  Quality of Life

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided